CLINICAL TRIAL: NCT04321577
Title: Prospective Validation of a Residual Disease Predictive Score in Incidental Gallbladder Cancer
Brief Title: Validation of a Score That Predicts Residual Disease in Incidental Gallbladder Cancer
Status: Withdrawn | Type: Observational
Why Stopped: At the beginning of the study, the collaboration of several Spanish liver surgery groups was planned. However, neither group has included a valid record. Likewise, the number of patients studied in our center has been extremely low.
Sponsor: Emilio Ramos (Other)
Responsible Party: Sponsor-Investigator, Emilio Ramos, Medical doctor, PhD, head of hepatic surgery, university professor, Hospital Universitari de Bellvitge
Organization: Hospital Universitari de Bellvitge (Other)
Other Study IDs: PR357/19
Record Dates: First submitted 2020-03-13; First posted 2020-03-25 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2020-07

CONDITIONS: Gallbladder Neoplasm Malignant Primary
Keywords: Residual disease; Risk score
MeSH Terms: conditions — Neoplasm, Residual

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples Without DNA — Cholecystectomy and re-resection specimen. Both of the fixed, sliced with a microtome in sections and stained with hematoxylin-eosin at the Pathology Laboratory.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Residual disease: Participants with incidental gallbladder cancer with presence of residual disease in the re-resection specimen or in intra-operative findings.
  Interventions: Procedure: Radical surgery
- No residual disease: Participants with incidental gallbladder cancer with absence of residual disease in the re-resection specimen or in intra-operative findings.
  Interventions: Procedure: Radical surgery

INTERVENTIONS:
Procedure: Radical surgery — Radical surgery is proposed to participants with pT1b, pT2 or pT3 tumors in the cholecystectomy specimen without evidence of disseminated disease with staging imaging techniques. A resection of the gallbladder bed or an anatomic resection of the hepatic segments IVb/V is performed. A lymphadenectomy of the hepatic hilum is associated in all cases. Common bile duct resection is performed in patients with involvement of the cystic margin.

SUMMARY:
An incidental gallbladder carcinoma is detected in approximately 0.2% of the cholecystectomy specimens removed for presumed benign disease. In patients that meet specific criteria, a surgical re-operation is recommended to treat possible residual tumor disease not treated with the initial cholecystectomy. The presence of residual disease in the re-intervention specimen worsens the prognosis of patient survival, according to several published series. Patients with known or high-risk of residual disease may benefit from a specific strategy that would improve patient selection before attempting re-resection. A pathology-based score has been developed but has not been yet validated in an external series of patients. The use of pathological data from the initial cholecystectomy specimen could identify patients at risk of residual disease and aid in selecting a specific therapeutic strategy prior to attempting surgical re-exploration.

DETAILED DESCRIPTION:
* Sample size: 30 (minimum).
* Statistical analysis: populations will be compared with chi-square test or Fisher's exact test (categorical variables) and Student's t test or Mann-Whitney U test (continuous variables). A univariate and multivariate logistic regression analysis will be performed to evaluate the predictive factors of residual disease. The Kaplan-Meier method will be applied for survival analysis and curves will be compared using log-rank test. Univariate and multivariate Cox proportional hazards ratio will be applied to determine the predictive factors of survival. Variables with p values inferior to 0.1 in the univariate analysis will be used to perform the multivariate analysis. Statistical significance is defined when p < 0.5. The statistical program used will be SPSS version 23.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients with a diagnosis of incidental gallbladder cancer requesting therapeutic evaluation in the participating hospital centers.

Exclusion Criteria:

* All patients with non-incidental gallbladder cancer.
* All patients with incomplete or deficient data collection.
* Patients without a signed informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with diagnosis of incidental gallbladder cancer that request therapeutic evaluation in the participating hospital centers.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-03 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Residual disease | Immediately after surgery in operated patients / within 1 year in non-operated patients
  Presence of tumoral cells in the re-resection specimen or found on staging imaging techniques. It can be local (isolated non-discontinuous involvement of the vesicular bed or the cystic stump), regional (common bile duct involvement, perineural, lymph node or neighboring organ invasion), or distant (discontinuous hepatic involvement -i.e. metastases-, peritoneal carcinomatosis or port-site metastases).
Gallbladder cancer risk score | Baseline
  Pathology-based score that uses T stage, grade of differentiation, presence of lymphovascular and perineural invasion evaluated in the cholecystectomy specimen to pre-operatively predict the presence of residual disease after radical resection. Each factor is assigned a value. Adding these values results in a total risk score that ranges between 3 and 10 points. The scores are separated intro three risk groups: low (3-4), intermediate (5-7) and high (8-10).

SECONDARY OUTCOMES:
Disease-specific survival | 1, 3, and 5-year disease-specific survival.
  Interval between date of surgical re-exploration and date of last follow-up or death. Only death from cancer will be considered an event in the analysis. Non-cancer related deaths will be excluded from the analysis.
Disease-free survival | 1, 3, and 5-year disease-free survival.
  Interval between date of surgical re-exploration and date of recurrence diagnosis (clinic, radiologic or pathologic) or last follow-up or death in patients without recurrence.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Lladó, MD, PhD, Principal Investigator — Hospital Universitari Bellvitge; Kristel Mills Julià, MD, Principal Investigator — Hospital Universitari Bellvitge
Locations (1):
- Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ramos E, Lluis N, Llado L, Torras J, Busquets J, Rafecas A, Serrano T, Mils K, Leiva D, Fabregat J. Prognostic value and risk stratification of residual disease in patients with incidental gallbladder cancer. World J Surg Oncol. 2020 Jan 24;18(1):18. doi: 10.1186/s12957-020-1794-2. PMID 31980034
- See also: Direct link to the previously cited article. — http://www.ncbi.nlm.nih.gov/pubmed/31980034